CLINICAL TRIAL: NCT03639662
Title: Psychological Impact of a Sophrological Accompaniment During the Announcement of Thyroid Cancer Compared With Usual Initial Management: Multicenter Randomized Prospective Study
Brief Title: Psychological Impact of a Sophrological Accompaniment During the Announcement of Thyroid Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RCAPHM18_0016
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Follicular Thyroid Cancer
MeSH Terms: conditions — Adenocarcinoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Patients benefit from additional support consisting of at least 3 sessions of sophrology (sophrology sessions), one per week, from the week following the announcement of the diagnosis and until the week preceding the hospitalization for "iratherapie". It will be group sessions, 1h carried out in the participating center by a nurse sophrologist who will use the techniques of sophrology such as relaxation, breath control, mastery of thoughts and visualization. Each session will be recorded in digital format and the recording will be given to the patient at the end of the session so that he can, if he wishes, reproduce it at home.
  Patients will also be able to share their feelings and ask questions
  Interventions: Other: sophrology sessions
- control group (No Intervention): Between the announcement of their thyroid cancer and the post-therapeutic scintigraphy, the patients will follow the usual route: information on the management, receipt of an information booklet (containing the telephone contacts of the hospital units), and they wish it, meet with the staff and visit a room of hospitalization. The nurses of the hospitalization service are available to answer any questions they may have, either during this visit or during a telephone call

INTERVENTIONS:
Other: sophrology sessions — Patients benefit from additional support consisting of at least 3 sessions of sophrology, one per week, from the week following the announcement of the diagnosis and until the week preceding the hospitalization for irathérapie. It will be group sessions, 1h carried out in the participating center by a nurse sophrologist who will use the techniques of sophrology such as relaxation, breath control, mastery of thoughts and visualization. Each session will be recorded in digital format and the recording will be given to the patient at the end of the session so that he can, if he wishes, reproduce it at home.
  Patients will also be able to share their feelings and ask questions
  Arms: experimental group

SUMMARY:
Follicular thyroid cancers are excellent prognoses. However, there is a very clear negative impact of the diagnosis on patients' quality of life, partly because of initial care. The therapeutic sequence is often the following: surgery and complementary administration of radioactive iodine 131. This treatment will destroy all thyroid cells remaining and thus minimize the risk of recurrence and facilitate future controls.

Radioactive iodine uptake is optimized by stimulating thyroid cells that fix iodine better when the level of TSH is high. For this purpose, hypothyroidism is induced by weaning in hormone replacement therapy or injected with recombinant TSH.

Then, a full-body scintigraphy extension is performed followed by a medical consultation. This scintigraphy shows the tissues that fixed the iodine 131, the residual tissues after surgery and / or possible distant metastases.

It is recognized that when a patient learns that he has thyroid cancer, he is subject to increasing anxiety between the time of diagnosis and post-treatment scintigraphy. These patients and their loved ones are often distraught and anticipate their future in a negative way, while long-term survival is excellent. How to get these patients to consider their pathology more objectively and thus reduce their anxiety?

Sophrology is a psychocorporal method aimed at balancing our emotions, thoughts and behaviors. We suppose that if these patients could benefit from a sophrological accompaniment between the announcement of the diagnosis and the scintigraphy, they could apprehend their pathology with more serenity and reality.

No studies providing sophrological support to patients with thyroid cancer have been performed. The anxiety of these patients being largely linked to a feeling of isolation and excessive danger, we think that this care will have an immediate favorable effect on their anxiety, or even in the longer term on their quality of life.

The aim is to offer patients a sophrological support provided by each of the 3 participating centers. These group sessions will allow them to understand the place of their future hospitalization, to share with other patients, to obtain answers to their questions, to be listened to with neutrality and empathy, and to learn management techniques. their anxiety in order to reproduce them at home. They will be followed and will not feel abandoned in the face of their distress.

DETAILED DESCRIPTION:
Follicular thyroid cancers are excellent prognoses (> 90% survival at all stages at 10 years). They occur preferentially in women where they represent the 5th cause of cancer and less than 0.5% of the causes of cancer mortality. However, there is a very clear negative impact of the diagnosis on patients' quality of life, partly because of initial care. The therapeutic sequence is often the following: surgery and complementary administration of radioactive iodine 131. This treatment will destroy all thyroid cells (normal or cancerous) remaining and thus minimize the risk of recurrence and facilitate future controls (the blood test of thyroglobulin produced only by the thyroid cells can be used as a marker of persistence / recurrence of the disease).

Radioactive iodine uptake is optimized by stimulating thyroid cells that fix iodine better when the level of TSH is high. For this purpose, hypothyroidism is induced by weaning in hormone replacement therapy or injected with recombinant TSH.

Approximately one week after iodine-131, a full-body scintigraphy extension is performed followed by a medical consultation. This scintigraphy shows the tissues that fixed the iodine 131, the residual tissues after surgery and / or possible distant metastases.

It is recognized that when a patient learns that he has thyroid cancer, he is subject to increasing anxiety between the time of diagnosis and post-treatment scintigraphy. These patients and their loved ones are often distraught and anticipate their future in a negative way, while long-term survival is excellent. How to get these patients to consider their pathology more objectively and thus reduce their anxiety?

Sophrology is a psychocorporal method aimed at balancing our emotions, thoughts and behaviors. We suppose that if these patients could benefit from a sophrological accompaniment between the announcement of the diagnosis and the scintigraphy, they could apprehend their pathology with more serenity and reality.

Previous work has already demonstrated the interest of sophrology in different situations such as the management of cancer patients, before performing a bronchial fibroscopy, a ventilation session as part of the management of cancer. neuropathic pain, but also in the elderly and finally in people cared for infertility.

No studies providing sophrological support to patients with thyroid cancer have been performed. The anxiety of these patients being largely linked to a feeling of isolation and excessive danger, we think that this care will have an immediate favorable effect on their anxiety, or even in the longer term on their quality of life.

The aim is to offer patients a sophrological support provided by each of the 3 participating centers (CHU Marseille, Institut Claudius Regaud Toulouse, Center Jean Perrin Clermont-Ferrand). These group sessions will allow them to understand the place of their future hospitalization, to share with other patients, to obtain answers to their questions, to be listened to with neutrality and empathy, and to learn management techniques. their anxiety in order to reproduce them at home. They will be followed and will not feel abandoned in the face of their distress.

ELIGIBILITY:
Inclusion Criteria:

* Major subject, affiliated to a social security scheme;
* Subject accepting to participate in the study and having signed informed consent; Subject with histologically confirmed follicular thyroid cancer (initial diagnosis);
* Subject having a minimum period of 4 weeks between surgery and the administration of iodine 131.

Exclusion Criteria:

Subjects with any of the following criteria will not be included:

* Subject with thyroid cancer known as distant metastatic
* Subject presenting another evolutionary cancer
* Subject not mastering the French language
* Subject presenting severe affective, behavioral or psychiatric disorders which, according to the investigator, compromise the ability to meet the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Score to STAI questionnaire | 1 hour
  The State-Trait Anxiety Inventory (STAI) is a self-questionnaire, developed by Spielberger (7) and validated in French. It has 20 questions, assessing the subject's usual emotional state. A score is calculated, ranging from 20 to 80, a high score indicating the presence of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France